CLINICAL TRIAL: NCT02627339
Title: A Prospective Study of Controls to Build a Normative Database for the Spaeth/Richman Contrast Sensitivity Test (SPARCS)
Brief Title: Building a Database of Results From People Without Eye Problems
Acronym: SPARCS
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Collaborators: Partridge Foundation (Unknown)
Responsible Party: Principal Investigator, George L. Spaeth MD, George L. Spaeth MD, Wills Eye
Other Study IDs: 12-234E
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: Contrast Sensitivity
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy controls: Healthy controls age 10 to 90 years

SUMMARY:
The purpose of this study is to build a database of results from a new test that measures contrast sensitivity (the Spaeth-Richman Contrast Sensitivity Test (SPARCS)). Contrast sensitivity is an important part of your ability to see. When contrast sensitivity decreases, you are less able to see objects and detect motion. For instance, if you have decreased contrast sensitivity, you might be less able to read, see in the dark, drive, hit a ball, or walk safely. Decrease in contrast sensitivity leads to a decrease in quality of life.

DETAILED DESCRIPTION:
Objective: To build a normative database for the Spaeth / Richman Contrast Sensitivity Test (SPARCS).

Background: Patients with glaucoma have diminished contrast sensitivity. SPARCS is a novel test designed to determine the contrast threshold in the central 5 degrees of vision as well as each of the 4 peripheral quadrants (superotemporal, superonasal, inferotemporal, inferonasal). It is performed on a standard computer with at least 1024 x 768 monitor resolution. The correct testing distance is 50 cm away from the computer screen. Appropriate refractive correction is used. Testing is performed in a room with standardized lighting (85 cd / m2) and no windows in order to minimize glare and reflections. Testing is performed monocularly with the non-tested eye covered by an eye patch. The purpose of this study is to build a normative database for SPARCS.

Study Design: Cross sectional observational study.

Methods: Healthy volunteers will be recruited from the Wills Eye Institute after obtaining informed consent following the principles of the Helsinki Convention. Approximately 320 people free of ocular disease will be recruited to form a portion of the normative database for SPARCS. A goal of 20 subjects per decade of life (10-19, 20-29, 30-39, 40-49, 50-59, 60-69, 70-79, 80+) for both Caucasians and African Americans will be recruited. Other ethnicities will also be recruited, though without specific recruitment goals. Future study locations will help diversify the population of the normative database.

After agreeing to participate in the study, subjects will be assessed to determine if they qualify. Potential participants will be asked if they have any known eye diseases or decreased vision. Best-corrected monocular visual acuities will be assessed using an ETDRS visual acuity chart. A slit lamp examination will be performed to confirm good ocular health. Subjects will be excluded if they have any apparent ocular disease that affects visual acuity or visual function. For example, people with glaucoma, macular degeneration, or diabetic retinopathy will be excluded. Additional exclusion criteria includes: visual acuity 20/40 or worse; cataract grade 2 3+ or worse; posterior capsular opacity grade 2 3+ or worse; refractive error greater than +5 or -5 diopters; and incisional eye surgery within the prior 3 months.

After a person qualifies for the normative database, he or she will then take SPARCS. A trained technician will position the patient to the correct testing distance, check room lighting, and then explain the test. Subjects will be told to fixate on the central area and when ready, click the central area once with a computer mouse. Vertical dark bars will briefly appear in 1 of the 5 tested areas on the computer monitor. A subject will then move the mouse to the area the image appeared and click it once. When the subject is ready for the next image to appear, he or she will click again on the central area. Subjects are also instructed to guess where the image appeared if unsure. Vertical square waves of varying contrast levels will then continue to appear in a random pattern until threshold has been reached for each area. After the testing algorithm has been completed, the test will automatically end.

Each eye of an eligible subject will take the test twice after receiving instructions from a technician. The technician will remain in the testing room the first two times SPARCS is taken. A half hour later, the subject will then take SPARCS again without instructions from the technician and without the technician being present in the room.

The mean score and standard deviation of each area and the total score will be analyzed for age, gender, race, and lens status. Spearman correlations will be used to examine continuous variables and Kruskal-Wallis analysis for categorical measures. Test-retest repeatability will be assessed using the Coefficient of Repeatability and the Intraclass Correlation Coefficient.

ELIGIBILITY:
Inclusion Criteria:

* 10 years or older and healthy
* No eye diseases

Exclusion Criteria:

* Patients with glaucoma, macular degeneration, diabetic retinopathy, corneal disease, eye movement disorders or any eye disease causing vision loss
* Patients with visual acuity worse than 20/40
* Patients with cataracts or opacities 2+ or greater
* Patients with refractive error +6 -6 or greater

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy controls with no eye diseases
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
SPARCS results | 1 day
  Results from each eyes response to the contrast sensitivity test

CONTACTS AND LOCATIONS:
Overall Officials: George L Spaeth, MD, Principal Investigator — Medical Director, Glaucoma Research Center
Locations (1):
- Wills Eye Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richman J, Spaeth GL, Wirostko B. Contrast sensitivity basics and a critique of currently available tests. J Cataract Refract Surg. 2013 Jul;39(7):1100-6. doi: 10.1016/j.jcrs.2013.05.001. Epub 2013 May 23. PMID 23706926